CLINICAL TRIAL: NCT03847025
Title: The Oregon Health & Science University Cardiac Implantable Electronic Device Extraction Registry
Brief Title: Pacemaker and Defibrillator Lead Extraction Registry
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Charles Henrikson, MD, Associate Professor of Medicine, Oregon Health and Science University
Other Study IDs: ER-9722
Record Dates: First submitted 2013-09-25; First posted 2019-02-20 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Lead Extraction Procedures
Keywords: Pacemaker; Implantable cardioverter defibrillator; Lead extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lead extraction: Patients undergoing clinically indicated lead extraction procedures.

SUMMARY:
Implanted cardiac devices are commonly used to treat a wide variety of heart diseases, including arrhythmias, cardiac resynchronization in select heart failure patients, and life threatening heart rhythms. Approximately 400,000 devices are implanted annually, and more than 3 million patients currently have implanted devices1.

Implanted cardiac devices are made to 2 components, the can and the leads. The can contains the electric circuits and the battery, which must be replaced every 5-10 years. The can is connected to external leads which pass through the subclavian vein, and depending on the device, into the vena cava, right atrium, right ventricle, and/or coronary sinus. Leads typically last longer than the battery, and are simply reconnected to a new can at the time of replacement.

Certain clinical situations necessitate lead removal, including pocket infection, device related endocarditis, venous stenosis or occlusion with the need for new access, and removal of abandoned or malfunctioning leads. Removing the leads is technically difficult due to fibrosis, and requires specialized equipment. Compared to lead implantation, extraction of leads is relatively rare, with a life time risk of a device patient needing an extraction in the 1-5% range. Given that this is a relatively rare procedure and is only done at a few centers, documentation of our experiences with lead extraction can lead to ongoing improvements in both procedural techniques and outcomes.

DETAILED DESCRIPTION:
Study Procedures

This is a retrospective review of data on patient characteristics (such as age, gender, co-morbidities), procedure specifications and indications, and outcomes of lead extraction done at OHSU.

Patients who have undergone either pacemaker or defibrillator lead extraction will have their charts reviewed for the desired data, which will then be compiled into a database. All procedures will be part of routine clinical care.

Data Analysis:

This is an observational registry study; there are no primary or secondary outcomes. Data will be analyzed to determine patient and procedural characteristics, procedure indications, complications and outcomes

ELIGIBILITY:
Inclusion Criteria:

- Undergoing lead extraction

Exclusion Criteria:

* registry--n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing clinically indicated lead extraction.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-09; Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
safety (acute complications, per HRS consensus document) | duration of hospitalization, typically 2 days to 2 weeks
  Primary outcome is safety of the lead extraction procedure, in terms of acute complications, per HRS consensus document.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Henrikson, MD, Principal Investigator — 503-494-0331
Locations (1):
- Charles Henrikson, Portland, Oregon, United States